CLINICAL TRIAL: NCT00378612
Title: Approaches to Chronic Occlusions With Sirolimus Stents-Cypher (ACROSS-Cypher) Total Occlusion Study of Coronary Arteries 4 Trial
Brief Title: ACROSS-Cypher Total Occlusion Study of Coronary Arteries 4 Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sunil Rao (Other)
Collaborators: Cordis US Corp. (Industry)
Responsible Party: Sponsor-Investigator, Sunil Rao, Associate Professor, Medicine - Cardiology, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00007965; 1525004 (Other: Legacy ID)
Record Dates: First submitted 2006-09-19; First posted 2006-09-20 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Coronary Occlusions
Keywords: trials; stents; coronary occlusions
MeSH Terms: conditions — Coronary Occlusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cypher® sirolimus eluting coronary stent (Experimental): All pts were given the Cypher sirolimus eluting coronary stent in this open-label, single-arm, non-randomized trial
  Interventions: Device: Cypher sirolimus eluting coronary stent

INTERVENTIONS:
Device: Cypher sirolimus eluting coronary stent — Cypher® sirolimus eluting coronary stent ranging in diameters 2.5 to 3.5 mm and available in length from 8 to 33 mm.

SUMMARY:
ACROSS-Cypher® is a prospective, multi-center, open label, single arm study of the Cypher® sirolimus eluting coronary stent in native total coronary occlusion revascularization. The primary endpoint is binary angiographic restenosis at 6 months. The TOSCA-1 trial will be used as the historical control. The hypothesis is that compared with TOSCA-1 patients who were treated with the heparin-coated Palmaz Schatz stent, treatment with the Cypher® sirolimus eluting coronary stent will result in a >50% relative reduction in 6 month restenosis within the treated segment of the target vessel.

DETAILED DESCRIPTION:
Despite remarkable advances in the procedural and clinical outcomes of percutaneous revascularization, chronically occluded coronary arteries remain a formidable challenge and unresolved dilemma in interventional cardiology. Although a TCO is identified in approximately one-third of diagnostic cardiac catheterizations, still an attempted revascularization accounts for less than 8% of all percutaneous coronary interventions (PCI). Such a disparity between their frequency and treatment not only underscores the technical and procedural frustrations associated with these complex lesions, but also the clinical uncertainties regarding clinical benefits with conventional TCO revascularization and the ongoing inadequacies of current PCI methods for sustaining restenosis-free patency following initial success.

Until recently, few clinical investigations have been performed to support clinical benefit of TCO revascularization. In addition to relief of symptomatic ischemia, theoretical advantages have included enhanced left ventricular function, reduced predisposition to arrhythmic events, and improved tolerance of future ischemic events. In the Survival and Ventricular Enlargement (SAVE) trial, persistent occlusion of the infarct-related artery was associated with a relative risk of 1.47 in adjusted 4-year mortality (P=0.04). Since then, a limited number of studies documenting long-term outcomes following intended TCO revascularization have been performed.

This investigational protocol is designed to evaluate the safety and efficacy of the Cypher® sirolimus eluting coronary stent (Cordis Corporation, Miami Lakes, FL) in patients undergoing elective revascularization of nonacute total coronary occlusions (TCO). Specifically, approximately 200 patients will undergo Cypher® sirolimus eluting coronary stent(s) implantation following successful crossing of native total occlusions with a coronary guidewire. The study will be conducted at approximately 17 sites in North America. Patients included in this trial will be scheduled for percutaneous revascularization of a non-acute de novo TCO in a native vessel visually estimated to accommodate a ≥3.0 mm diameter angioplasty balloon. Important exclusion criteria will include recent myocardial infarction (<72 hours) and any general contraindication to the procedure or scheduled clinical and angiographic follow-up. Patients may also undergo treatment of a non-target vessel lesion simultaneous with the index procedure within certain protocol-specified provisions. All patients will undergo planned angiographic follow-up 6 months following the index procedure to evaluate the primary endpoint of restenosis (>50% diameter stenosis) within the treated/working length segment compared with results obtained using the same methodology among patients undergoing TCO revascularization with the heparin-coated Palmaz-Schatz coronary stent (Cordis Corporation, Miami Lakes, FL) in the Total Occlusion Study of Canada-1 (TOSCA) (1). Important secondary endpoints include the occurrence of major adverse cardiac events (MACE) and target vessel failure (TVF) at 30 days, 6 months and 12 months post-procedure. In addition, angiographic outcomes of in-stent and segment restenosis within the stent and segment will be examined. Further, patients enrolled in the trial will have clinical follow-up annually to five years.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 years or older at time of consent
* Patients with clinical symptoms suggesting ischemic heart disease or having evidence of myocardial ischemia and scheduled for clinically indicated percutaneous revascularization
* Eligibility and consent to undergo PCI procedure
* Patient is an acceptable candidate for percutaneous transluminal coronary angioplasty,stenting,and emergency coronary artery bypass grafting
* Willing and able to sign informed consent form approved by local IRB/Ethics Committee and to follow protocol, including 6-month follow-up angiography
* At least 1 target segment meeting definition of non-acute total coronary occlusion
* High-grade native coronary stenosis
* Thrombolysis in Myocardial Infarction 0 or 1 antegrade flow
* Target occlusion successfully crossed with commercially available coronary guidewire
* Occluded segment suitable for placement of coronary stents
* Treated segment can accommodate 3.0mm or greater diameter balloon
* Segment not beyond severe tortuosity (45° or more) or excessively distal location

Exclusion Criteria:

* Patients undergoing treatment of a non-target vessel that is also a total coronary occlusion
* Patients with any history of allergy to iodinated contrast that cannot be effectively managed medically, or any known allergy to clopidogrel bisulfate (Plavix®), aspirin, heparin, ticlopidine, stainless steel, or sirolimus
* Evidence of acute myocardial infarction within 72 hours of intended treatment (Q-wave or non-Q-wave myocardial infarction having creatine kinase enzymes 2X the upper limit of normal with presence of a creatine kinase myocardial-band isoenzyme above Institution's ULN, or troponin above the Institution's ULN)
* Previous coronary interventional procedure of any kind within 3 months prior to the procedure in target vessel
* Planned interventional treatment of either target or any non-target vessel within 30 days post-procedure with a bare metal or Cypher® sirolimus eluting coronary stent
* Planned interventional treatment of either the target or any non-target vessel within 6 months post-procedure with a paclitaxel-eluting TAXUSTM stent
* Any contraindication to cardiac catheterization or to any standard concomitant therapies used during routine cardiac catheterization and PCI
* Target lesion requires planned treatment with a device after successful crossing other than PTCA prior to stent
* Patients with history of clinically significant abnormal laboratory findings including
* Current (within previous two weeks) neutropenia (<1000 neutrophils/mm3)
* Thrombocytopenia (<100,000 platelets/mm3)
* AST, ALT, alkaline phosphatase, or bilirubin > 1.5XULN
* Serum creatinine > 1.5 mg/dL
* Patients with evidence of ongoing or active clinical instability including the following
* Sustained systolic blood pressure < 100mmHg or cardiogenic shock
* Acute pulmonary edema or severe congestive heart failure
* Suspected acute myocarditis, pericarditis, endocarditis, or cardiac tamponade
* Suspected dissecting aortic aneurysm
* Hemodynamically significant valvular heart disease, hypertrophic cardiomyopathy, restrictive cardiomyopathy, or congenital heart disease
* Target lesion involves a bifurcation including a diseased side branch 2.25mm or more in diameter requiring treatment
* Prior coronary bypass surgery of target lesion with patent bypass graft (balloon angioplasty alone, without coronary stenting, is permitted)
* History of stroke or transient ischemic attack within prior 6 months
* Female patients of childbearing potential
* Active peptic ulcer or upper gastrointestinal bleeding within prior 6 months
* History of bleeding diathesis or coagulopathy or refusal of blood transfusions
* Patients with any other pathology such as cancer, mental illness, which in the opinion of the investigator, might put the patient at risk, preclude follow-up, or in any way confound the results of the study
* Known previous medical condition yielding expected survival less than 1 year
* Patients who are unable or unwilling to comply with the protocol or not expected to complete the study period, including its follow-up requirements
* Currently participating in an investigational drug or another device study that has not completed the primary endpoint or that clinically interferes with the current study endpoints; or requires coronary angiography, intravascular ultrasound, or other coronary artery imaging procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2005-06; Primary Completion 2007-04 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Angiographic binary restenosis (>=50% diameter stenosis) in TCO treated/working length compared with restenosis outcomes in the Total Occlusion Study of Canada (TOSCA) | 6 months post-procedure

SECONDARY OUTCOMES:
Angiographic binary in-segment restenosis (>= 50% diameter stenosis) rate at 6 months post-procedure | 6 months post-procedure
Angiographic binary in-stent restenosis (>= 50% diameter stenosis) rate at 6 months post-procedure | 6 months post-procedure
In-segment late lumen loss at 6 months | 6 months post-procedure
In-stent late lumen loss at 6 months | 6 months post-procedure
Device Success | 6 months post-procedure
Lesion Success | 6 months post-procedure
Procedure Success | 6 months post-procedure
Major Adverse Cardiac Events (MACE) rate at 30 days, 6 months, and 12 months post-procedure | 30 days, 6 months and 12 months post-procedure
Target Site Revascularization (TSR) rate and clinically-driven TSR rate at 6 and 12 months post-procedure Target Vessel Revascularization (TVR) rate and clinically-driven TVR rate at 6 and 12 months post-procedure | 6 and 12 months post-procedure
Target Vessel Failure (TVF) rate at 6 and 12 months post-procedure | 6 and 12 months post-procedure
In-stent and in-segment minimum lumen diameter (MLD) at 6 months post-procedure | 6 months post-procedure
Failure of sustained patency at 6 months (≥70% stenosis with TIMI <3 flow at follow-up angiography) | 6 months post-procedure
Subacute thrombosis occurring within 30 days post-procedure | 30 days post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Rao, M.D., Principal Investigator — Duke University
Locations (16):
- United States (13):
  - Green Hospital of Scripps Health, La Jolla, California
  - Scripps Memorial Hospital-La Jolla, La Jolla, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Emory University, Atlanta, Georgia
  - Brigham and Womens Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - William Beaumont Hospital, Royal Oak, Michigan
  - Saint Lukes Hospital, Kansas City, Missouri
  - New York Presbyterian Medical, New York, New York
  - The Sanger Clinic PA, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - North Ohio Heart Center, Elyria, Ohio
  - Heart Hospital of Austin, Austin, Texas
- Canada (3):
  - Vancouver Hospital and Health Science Centre, Vancouver, British Columbia
  - Saint Michaels Hospital, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario

REFERENCES:
- [Background] Buller CE, Dzavik V, Carere RG, Mancini GB, Barbeau G, Lazzam C, Anderson TJ, Knudtson ML, Marquis JF, Suzuki T, Cohen EA, Fox RS, Teo KK. Primary stenting versus balloon angioplasty in occluded coronary arteries: the Total Occlusion Study of Canada (TOSCA). Circulation. 1999 Jul 20;100(3):236-42. doi: 10.1161/01.cir.100.3.236. PMID 10411846
- [Background] Srinivas VS, Brooks MM, Detre KM, King SB 3rd, Jacobs AK, Johnston J, Williams DO. Contemporary percutaneous coronary intervention versus balloon angioplasty for multivessel coronary artery disease: a comparison of the National Heart, Lung and Blood Institute Dynamic Registry and the Bypass Angioplasty Revascularization Investigation (BARI) study. Circulation. 2002 Sep 24;106(13):1627-33. doi: 10.1161/01.cir.0000031570.27023.79. PMID 12270854
- [Background] Noguchi T, Miyazaki MD S, Morii I, Daikoku S, Goto Y, Nonogi H. Percutaneous transluminal coronary angioplasty of chronic total occlusions. Determinants of primary success and long-term clinical outcome. Catheter Cardiovasc Interv. 2000 Mar;49(3):258-64. doi: 10.1002/(sici)1522-726x(200003)49:33.0.co;2-l. PMID 10700054
- [Background] Ivanhoe RJ, Weintraub WS, Douglas JS Jr, Lembo NJ, Furman M, Gershony G, Cohen CL, King SB 3rd. Percutaneous transluminal coronary angioplasty of chronic total occlusions. Primary success, restenosis, and long-term clinical follow-up. Circulation. 1992 Jan;85(1):106-15. doi: 10.1161/01.cir.85.1.106. PMID 1728439
- [Background] Lamas GA, Flaker GC, Mitchell G, Smith SC Jr, Gersh BJ, Wun CC, Moye L, Rouleau JL, Rutherford JD, Pfeffer MA, et al. Effect of infarct artery patency on prognosis after acute myocardial infarction. The Survival and Ventricular Enlargement Investigators. Circulation. 1995 Sep 1;92(5):1101-9. doi: 10.1161/01.cir.92.5.1101. PMID 7648653
- [Background] Suero JA, Marso SP, Jones PG, Laster SB, Huber KC, Giorgi LV, Johnson WL, Rutherford BD. Procedural outcomes and long-term survival among patients undergoing percutaneous coronary intervention of a chronic total occlusion in native coronary arteries: a 20-year experience. J Am Coll Cardiol. 2001 Aug;38(2):409-14. doi: 10.1016/s0735-1097(01)01349-3. PMID 11499731
- [Background] Farr AD. Letter: Status of medical laboratory scientists. Br Med J. 1976 Jun 19;1(6024):1534. doi: 10.1136/bmj.1.6024.1534-d. No abstract available. PMID 1276764
- [Background] Maiello L, Colombo A, Gianrossi R, Mutinelli MR, Bouzon R, Thomas J, Finci L. Coronary angioplasty of chronic occlusions: factors predictive of procedural success. Am Heart J. 1992 Sep;124(3):581-4. doi: 10.1016/0002-8703(92)90262-t. PMID 1514482
- [Background] Sirnes PA, Golf S, Myreng Y, Molstad P, Emanuelsson H, Albertsson P, Brekke M, Mangschau A, Endresen K, Kjekshus J. Stenting in Chronic Coronary Occlusion (SICCO): a randomized, controlled trial of adding stent implantation after successful angioplasty. J Am Coll Cardiol. 1996 Nov 15;28(6):1444-51. doi: 10.1016/s0735-1097(96)00349-x. PMID 8917256
- [Background] Hoher M, Wohrle J, Grebe OC, Kochs M, Osterhues HH, Hombach V, Buchwald AB. A randomized trial of elective stenting after balloon recanalization of chronic total occlusions. J Am Coll Cardiol. 1999 Sep;34(3):722-9. doi: 10.1016/s0735-1097(99)00254-5. PMID 10483953
- [Background] Rubartelli P, Niccoli L, Verna E, Giachero C, Zimarino M, Fontanelli A, Vassanelli C, Campolo L, Martuscelli E, Tommasini G. Stent implantation versus balloon angioplasty in chronic coronary occlusions: results from the GISSOC trial. Gruppo Italiano di Studio sullo Stent nelle Occlusioni Coronariche. J Am Coll Cardiol. 1998 Jul;32(1):90-6. doi: 10.1016/s0735-1097(98)00193-4. PMID 9669254
- [Background] Mori M, Kurogane H, Hayashi T, Yasaka Y, Ohta S, Kajiya T, Takarada A, Yoshida A, Matsuda Y, Nakagawa K, Murata T, Yoshida Y, Yokoyama M. Comparison of results of intracoronary implantation of the Plamaz-Schatz stent with conventional balloon angioplasty in chronic total coronary arterial occlusion. Am J Cardiol. 1996 Nov 1;78(9):985-9. doi: 10.1016/s0002-9149(96)00521-8. PMID 8916475
- [Background] Lotan C, Rozenman Y, Hendler A, Turgeman Y, Ayzenberg O, Beyar R, Krakover R, Rosenfeld T, Gotsman MS. Stents in total occlusion for restenosis prevention. The multicentre randomized STOP study. The Israeli Working Group for Interventional Cardiology. Eur Heart J. 2000 Dec;21(23):1960-6. doi: 10.1053/euhj.2000.2295. PMID 11071802
- [Background] Sedel'nikov GN. [Friendship and cooperation]. Voen Med Zh. 1976 Mar;(3):78-81. No abstract available. Russian. PMID 1274228
- [Background] Sirnes PA, Golf S, Myreng Y, Molstad P, Albertsson P, Mangschau A, Endresen K, Kjekshus J. Sustained benefit of stenting chronic coronary occlusion: long-term clinical follow-up of the Stenting in Chronic Coronary Occlusion (SICCO) study. J Am Coll Cardiol. 1998 Aug;32(2):305-10. doi: 10.1016/s0735-1097(98)00247-2. PMID 9708454
- [Background] Serruys PW, de Jaegere P, Kiemeneij F, Macaya C, Rutsch W, Heyndrickx G, Emanuelsson H, Marco J, Legrand V, Materne P, et al. A comparison of balloon-expandable-stent implantation with balloon angioplasty in patients with coronary artery disease. Benestent Study Group. N Engl J Med. 1994 Aug 25;331(8):489-95. doi: 10.1056/NEJM199408253310801. PMID 8041413
- [Background] Moses JW, Leon MB, Popma JJ, Fitzgerald PJ, Holmes DR, O'Shaughnessy C, Caputo RP, Kereiakes DJ, Williams DO, Teirstein PS, Jaeger JL, Kuntz RE; SIRIUS Investigators. Sirolimus-eluting stents versus standard stents in patients with stenosis in a native coronary artery. N Engl J Med. 2003 Oct 2;349(14):1315-23. doi: 10.1056/NEJMoa035071. PMID 14523139
- [Background] Hoye A, Tanabe K, Lemos PA, Aoki J, Saia F, Arampatzis C, Degertekin M, Hofma SH, Sianos G, McFadden E, van der Giessen WJ, Smits PC, de Feyter PJ, van Domburg RT, Serruys PW. Significant reduction in restenosis after the use of sirolimus-eluting stents in the treatment of chronic total occlusions. J Am Coll Cardiol. 2004 Jun 2;43(11):1954-8. doi: 10.1016/j.jacc.2004.01.045. PMID 15172397
- [Background] Nakamura S, Muthusamy TS, Bae JH, Cahyadi YH, Udayachalerm W, Tresukosol D. Impact of sirolimus-eluting stent on the outcome of patients with chronic total occlusions. Am J Cardiol. 2005 Jan 15;95(2):161-6. doi: 10.1016/j.amjcard.2004.08.088. PMID 15642545
- [Background] Werner GS, Krack A, Schwarz G, Prochnau D, Betge S, Figulla HR. Prevention of lesion recurrence in chronic total coronary occlusions by paclitaxel-eluting stents. J Am Coll Cardiol. 2004 Dec 21;44(12):2301-6. doi: 10.1016/j.jacc.2004.09.040. PMID 15607390
- [Background] Waksman R, Robinson KA, Crocker IR, Wang C, Gravanis MB, Cipolla GD, Hillstead RA, King SB 3rd. Intracoronary low-dose beta-irradiation inhibits neointima formation after coronary artery balloon injury in the swine restenosis model. Circulation. 1995 Nov 15;92(10):3025-31. doi: 10.1161/01.cir.92.10.3025. PMID 7586273
- [Background] Wiedermann JG, Marboe C, Amols H, Schwartz A, Weinberger J. Intracoronary irradiation markedly reduces neointimal proliferation after balloon angioplasty in swine: persistent benefit at 6-month follow-up. J Am Coll Cardiol. 1995 May;25(6):1451-6. doi: 10.1016/0735-1097(95)00010-2. PMID 7722148
- [Background] Verin V, Popowski Y, Urban P, Belenger J, Redard M, Costa M, Widmer MC, Rouzaud M, Nouet P, Grob E, et al. Intra-arterial beta irradiation prevents neointimal hyperplasia in a hypercholesterolemic rabbit restenosis model. Circulation. 1995 Oct 15;92(8):2284-90. doi: 10.1161/01.cir.92.8.2284. PMID 7554213
- [Background] Wiedermann JG, Marboe C, Amols H, Schwartz A, Weinberger J. Intracoronary irradiation markedly reduces restenosis after balloon angioplasty in a porcine model. J Am Coll Cardiol. 1994 May;23(6):1491-8. doi: 10.1016/0735-1097(94)90397-2. PMID 8176112
- [Background] Faxon DP, Spiro TE, Minor S, Cote G, Douglas J, Gottlieb R, Califf R, Dorosti K, Topol E, Gordon JB, et al. Low molecular weight heparin in prevention of restenosis after angioplasty. Results of Enoxaparin Restenosis (ERA) Trial. Circulation. 1994 Aug;90(2):908-14. doi: 10.1161/01.cir.90.2.908. PMID 8044962
- [Background] Holmes DR Jr, Savage M, LaBlanche JM, Grip L, Serruys PW, Fitzgerald P, Fischman D, Goldberg S, Brinker JA, Zeiher AM, Shapiro LM, Willerson J, Davis BR, Ferguson JJ, Popma J, King SB 3rd, Lincoff AM, Tcheng JE, Chan R, Granett JR, Poland M. Results of Prevention of REStenosis with Tranilast and its Outcomes (PRESTO) trial. Circulation. 2002 Sep 3;106(10):1243-50. doi: 10.1161/01.cir.0000028335.31300.da. PMID 12208800
- [Background] Steinhubl SR, Berger PB, Mann JT 3rd, Fry ET, DeLago A, Wilmer C, Topol EJ; CREDO Investigators. Clopidogrel for the Reduction of Events During Observation. Early and sustained dual oral antiplatelet therapy following percutaneous coronary intervention: a randomized controlled trial. JAMA. 2002 Nov 20;288(19):2411-20. doi: 10.1001/jama.288.19.2411. PMID 12435254
- [Background] Kutryk MJ, Foley DP, van den Brand M, Hamburger JN, van der Giessen WJ, deFeyter PJ, Bruining N, Sabate M, Serruys PW; ITALICS Trial. Local intracoronary administration of antisense oligonucleotide against c-myc for the prevention of in-stent restenosis: results of the randomized investigation by the Thoraxcenter of antisense DNA using local delivery and IVUS after coronary stenting (ITALICS) trial. J Am Coll Cardiol. 2002 Jan 16;39(2):281-7. doi: 10.1016/s0735-1097(01)01741-7. PMID 11788220
- [Background] de Feyter PJ, Vos J, Rensing BJ. Anti-restenosis Trials. Curr Interv Cardiol Rep. 2000 Nov;2(4):326-331. PMID 11096683
- [Background] Marx SO, Jayaraman T, Go LO, Marks AR. Rapamycin-FKBP inhibits cell cycle regulators of proliferation in vascular smooth muscle cells. Circ Res. 1995 Mar;76(3):412-7. doi: 10.1161/01.res.76.3.412. PMID 7532117
- [Background] Mohacsi PJ, Tuller D, Hulliger B, Wijngaard PL. Different inhibitory effects of immunosuppressive drugs on human and rat aortic smooth muscle and endothelial cell proliferation stimulated by platelet-derived growth factor or endothelial cell growth factor. J Heart Lung Transplant. 1997 May;16(5):484-92. PMID 9171265
- [Background] Poon M, Marx SO, Gallo R, Badimon JJ, Taubman MB, Marks AR. Rapamycin inhibits vascular smooth muscle cell migration. J Clin Invest. 1996 Nov 15;98(10):2277-83. doi: 10.1172/JCI119038. PMID 8941644
- [Background] Burke SE, Lubbers NL, Chen YW, Hsieh GC, Mollison KW, Luly JR, Wegner CD. Neointimal formation after balloon-induced vascular injury in Yucatan minipigs is reduced by oral rapamycin. J Cardiovasc Pharmacol. 1999 Jun;33(6):829-35. doi: 10.1097/00005344-199906000-00001. PMID 10367584
- [Background] Gregory CR, Huang X, Pratt RE, Dzau VJ, Shorthouse R, Billingham ME, Morris RE. Treatment with rapamycin and mycophenolic acid reduces arterial intimal thickening produced by mechanical injury and allows endothelial replacement. Transplantation. 1995 Mar 15;59(5):655-61. doi: 10.1097/00007890-199503150-00002. PMID 7533955
- [Background] Gregory CR, Huie P, Billingham ME, Morris RE. Rapamycin inhibits arterial intimal thickening caused by both alloimmune and mechanical injury. Its effect on cellular, growth factor, and cytokine response in injured vessels. Transplantation. 1993 Jun;55(6):1409-18. doi: 10.1097/00007890-199306000-00037. PMID 8516827
- [Background] Poston RS, Billingham M, Hoyt EG, Pollard J, Shorthouse R, Morris RE, Robbins RC. Rapamycin reverses chronic graft vascular disease in a novel cardiac allograft model. Circulation. 1999 Jul 6;100(1):67-74. doi: 10.1161/01.cir.100.1.67. PMID 10393683
- [Background] Gallo R, Padurean A, Jayaraman T, Marx S, Roque M, Adelman S, Chesebro J, Fallon J, Fuster V, Marks A, Badimon JJ. Inhibition of intimal thickening after balloon angioplasty in porcine coronary arteries by targeting regulators of the cell cycle. Circulation. 1999 Apr 27;99(16):2164-70. doi: 10.1161/01.cir.99.16.2164. PMID 10217658
- [Background] Sousa JE, Costa MA, Abizaid A, Abizaid AS, Feres F, Pinto IM, Seixas AC, Staico R, Mattos LA, Sousa AG, Falotico R, Jaeger J, Popma JJ, Serruys PW. Lack of neointimal proliferation after implantation of sirolimus-coated stents in human coronary arteries: a quantitative coronary angiography and three-dimensional intravascular ultrasound study. Circulation. 2001 Jan 16;103(2):192-5. doi: 10.1161/01.cir.103.2.192. PMID 11208675
- [Background] Sousa JE, Costa MA, Abizaid AC, Rensing BJ, Abizaid AS, Tanajura LF, Kozuma K, Van Langenhove G, Sousa AG, Falotico R, Jaeger J, Popma JJ, Serruys PW. Sustained suppression of neointimal proliferation by sirolimus-eluting stents: one-year angiographic and intravascular ultrasound follow-up. Circulation. 2001 Oct 23;104(17):2007-11. doi: 10.1161/hc4201.098056. PMID 11673337
- [Background] Morice MC, Serruys PW, Sousa JE, Fajadet J, Ban Hayashi E, Perin M, Colombo A, Schuler G, Barragan P, Guagliumi G, Molnar F, Falotico R; RAVEL Study Group. Randomized Study with the Sirolimus-Coated Bx Velocity Balloon-Expandable Stent in the Treatment of Patients with de Novo Native Coronary Artery Lesions. A randomized comparison of a sirolimus-eluting stent with a standard stent for coronary revascularization. N Engl J Med. 2002 Jun 6;346(23):1773-80. doi: 10.1056/NEJMoa012843. PMID 12050336
- [Background] Sousa JE, Costa MA, Abizaid A, Sousa AG, Feres F, Mattos LA, Centemero M, Maldonado G, Abizaid AS, Pinto I, Falotico R, Jaeger J, Popma JJ, Serruys PW. Sirolimus-eluting stent for the treatment of in-stent restenosis: a quantitative coronary angiography and three-dimensional intravascular ultrasound study. Circulation. 2003 Jan 7;107(1):24-7. doi: 10.1161/01.cir.0000047063.22006.41. PMID 12515737
- [Background] Schampaert E, Cohen EA, Schluter M, Reeves F, Traboulsi M, Title LM, Kuntz RE, Popma JJ; C-SIRIUS Investigators. The Canadian study of the sirolimus-eluting stent in the treatment of patients with long de novo lesions in small native coronary arteries (C-SIRIUS). J Am Coll Cardiol. 2004 Mar 17;43(6):1110-5. doi: 10.1016/j.jacc.2004.01.024. PMID 15028375
- [Background] Colombo A, Moses JW, Morice MC, Ludwig J, Holmes DR Jr, Spanos V, Louvard Y, Desmedt B, Di Mario C, Leon MB. Randomized study to evaluate sirolimus-eluting stents implanted at coronary bifurcation lesions. Circulation. 2004 Mar 16;109(10):1244-9. doi: 10.1161/01.CIR.0000118474.71662.E3. Epub 2004 Feb 23. PMID 14981005
- [Background] Loginova EA, Potekhina MV, Khondkarian ShG, Korolev VS. [Specialization and rational use of hospital funds (based on materials of the city of Kalinin)]. Zdravookhr Ross Fed. 1976 Mar;(3):11-6. No abstract available. Russian. PMID 983430
- [Background] Robins JM, Hernan MA, Brumback B. Marginal structural models and causal inference in epidemiology. Epidemiology. 2000 Sep;11(5):550-60. doi: 10.1097/00001648-200009000-00011. PMID 10955408
- [Background] Stone GW, Ellis SG, Cox DA, Hermiller J, O'Shaughnessy C, Mann JT, Turco M, Caputo R, Bergin P, Greenberg J, Popma JJ, Russell ME; TAXUS-IV Investigators. A polymer-based, paclitaxel-eluting stent in patients with coronary artery disease. N Engl J Med. 2004 Jan 15;350(3):221-31. doi: 10.1056/NEJMoa032441. PMID 14724301
- [Background] Lunceford JK, Davidian M. Stratification and weighting via the propensity score in estimation of causal treatment effects: a comparative study. Stat Med. 2004 Oct 15;23(19):2937-60. doi: 10.1002/sim.1903. PMID 15351954
- [Background] D'Agostino RB Jr. Propensity score methods for bias reduction in the comparison of a treatment to a non-randomized control group. Stat Med. 1998 Oct 15;17(19):2265-81. doi: 10.1002/(sici)1097-0258(19981015)17:193.0.co;2-b. PMID 9802183
- [Result] Waksman R, Robinson KA, Crocker IR, Gravanis MB, Cipolla GD, King SB 3rd. Endovascular low-dose irradiation inhibits neointima formation after coronary artery balloon injury in swine. A possible role for radiation therapy in restenosis prevention. Circulation. 1995 Mar 1;91(5):1533-9. doi: 10.1161/01.cir.91.5.1533. PMID 7867195
- [Derived] Kandzari DE, Rao SV, Moses JW, Dzavik V, Strauss BH, Kutryk MJ, Simonton CA, Garg J, Lokhnygina Y, Mancini GB, Yeoh E, Buller CE; ACROSS/TOSCA-4 Investigators. Clinical and angiographic outcomes with sirolimus-eluting stents in total coronary occlusions: the ACROSS/TOSCA-4 (Approaches to Chronic Occlusions With Sirolimus-Eluting Stents/Total Occlusion Study of Coronary Arteries-4) trial. JACC Cardiovasc Interv. 2009 Feb;2(2):97-106. doi: 10.1016/j.jcin.2008.10.013. PMID 19463409